CLINICAL TRIAL: NCT02471937
Title: Integrative Approach to Identify Environmental Risk Factors for CC-17 Group B Streptococcal Neonatal Infection
Acronym: STREPB17
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2014-A01824-43
Record Dates: First submitted 2015-03-31; First posted 2015-06-15 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Vaginal Colonization With GBS
Keywords: Streptococcus agalactiae; Group B Streptococcus; Neonates; colonization; meningitis; Clonal Complex CC17; microbiota; next generation sequencing (NGS)
MeSH Terms: conditions — Meningitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregnant women negative for GBS colonization (Experimental): Only women negative for GBS during all the study will be included.
  Interventions: Biological: Bacteriological analyses on clinical samples performed with Eswabs

INTERVENTIONS:
Biological: Bacteriological analyses on clinical samples performed with Eswabs — Clinical samples analysed :
  mothervagina, breast milk, baby oral cavity, baby stool. Techniques: bacteriological cultures, Real time PCR

SUMMARY:
Streptococcus agalactiae (GBS) is the leading cause of neonatal septicaemia, meningitis, and pneumonia in the industrialized world. Early onset (EOD) and late onset (LOD) diseases are defined in neonates by their occurring within or after the first week of life, respectively. Molecular epidemiological studies have identified a capsular serotype III clone, referred to as CC-17 by Multi Locus Sequence Typing, as accounting for the vast majority of neonatal invasive diseases and for almost all cases of meningitis in LOD.

The investigators working hypothesis is that host-environmental interactions may contribute to the colonization and persistence of the hypervirulent CC-17 GBS in the neonate. In this project the investigators will determine if reciprocal interactions between the intestinal microbiota and the innate and adaptive immune system may specifically facilitate the colonization of the neonate by the hypervirulent GBS CC-17 clone.

DETAILED DESCRIPTION:
Four specific tasks will be addressed to:

(i) Understand whether and how the gut microbiota may influence growth and colonization of GBS CC-17 within the intestine of neonates.

(ii) Study the contribution of different diets and immune system constituents enabling the persistence of GBS CC-17 in the gut of neonates.

(iii) Determine whether the adaptive immune response elicited by maternal GBS colonization and transmitted to the infant is different for GBS CC-17 versus non-CC-17 GBS.

(iv) Determine whether or not GBS strains isolated from the mothers and from their babies are identical and whether the environment (ie. the vagina or the milk for the mother, the intestine or the oral cavity for the baby) influence the expression of specific virulence factors of CC-17.

ELIGIBILITY:
Inclusion criteria:

* Patient having a negative vaginal swab for GBS at 35-37 weeks
* Patient aged over 18 years
* Patient who received information and agreeing to sign informed consent
* Patient affiliated or beneficiary of an insurance

Exclusion criteria:

* Patient does not speak and does not understand French

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-04-28 (Actual); Study Completion 2016-04-28 (Actual)

PRIMARY OUTCOMES:
Number of Negative GBS screening in vaginal samples | 2 months

SECONDARY OUTCOMES:
Number of Negative GBS screening in fecal samples . | 2 months
Number of Negative GBS screening in fecal samples . | at birth
Number of Negative GBS screening in vaginal samples | At delivery

CONTACTS AND LOCATIONS:
Overall Officials: Claire POYART, MD, PhD,, Study Director — Assistance Publique Hôpitaux de Paris, Université Paris Descartes
Locations (1):
- CH Louis Mourier, Colombes, France

REFERENCES:
- [Background] Plainvert C, Anselem O, Joubrel C, Marcou V, Falloukh A, Frigo A, Magdoud El Alaoui F, Ancel PY, Jarreau PH, Mandelbrot L, Goffinet F, Poyart C, Tazi A. Persistence of group B Streptococcus vaginal colonization and prevalence of hypervirulent CC-17 clone correlate with the country of birth: a prospective 3-month follow-up cohort study. Eur J Clin Microbiol Infect Dis. 2021 Jan;40(1):133-140. doi: 10.1007/s10096-020-04011-6. Epub 2020 Aug 18. PMID 32812077